CLINICAL TRIAL: NCT05852171
Title: A Prospective Open-label Single-arm Clinical Study of the Efficacy of Baricitinib for Idiopathic Granulomatous Mastitis in a Single Institution
Brief Title: Baricitinib in Idiopathic Granulomatous Mastitis
Acronym: B-IGM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZYYY-IGM-001
Record Dates: First submitted 2023-04-23; First posted 2023-05-10 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-05

CONDITIONS: Mastitis Chronic; Idiopathic Granulomatous Mastitis
Keywords: Baricitinib
MeSH Terms: interventions — baricitinib

STUDY DESIGN:
Intervention Model Description: This study is a single-center, non-controlled, open-label, prospective single-arm trial (Simon's two-stage design). To evaluate the clinical efficacy and safety of baricitinib for idiopathic granulomatous mastitis. At least 20 patients are planned to be enrolled, and the objective response rate including clinical complete remission rate and partial response rate is the main endpoint.This study will also assess the degree of focus reduction, the recurrence rate within 12 months after drug termination, the degree of inflammation markers decline, and the toxicity and side effects of the drug.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Baricitinib (Experimental): Baricitinib，2mg QD，oral use.
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — Baricitinib administered orally
  Other Names: Olumiant; Baricinix

SUMMARY:
This study will explore the mechanism of targeted drug in treatment of idiopathic granulomatous mastitis, and clarify the clinical classification and corresponding markers.

DETAILED DESCRIPTION:
This study is aimed to explore the treatment effect of baricitinib in idiopathic granulomatous mastitis (IGM), as well as the clinical classification, potential markers and underline etiology of the disease. The target population of interest in this study is patients with non-lactating mastitis, which require core needle biopsy pathology to indicate mastitis without any pathogen infection. When IGM was diagnosed and informed consent complete, low dose of daily 2mg baricitinib was taken orally as the monotherapy in this trial. Follow-up visits were sheduled at baseline (i.e. pretreatment) , 1,3,6 months after treatment, and then every 3 months thereafter until 2 years after treatment discontinuation when achieving complete response. At each follow-up visit, the biggest IGM lesion in each patient was measured by breast ultrasound and 12 inflammational cytokines in peripheral blood should be tested. The primary end point was the objective response rate (ORR) including clinical complete response rate (CR) and partial response rate (PR), and the secondary end point was the recurrence rate within 12 months after drug discontinuation when achieving CR, the degree of inflammation markers decline, and the toxicity and side effects of the drug.

ELIGIBILITY:
[Inclusion Criteria]

Patients who are willing to participate in clinical research; females; age 18-70 years; KPS>80%, ECOG<2; non-lactating mastitis; core needle biopsy pathology suggests mastitis or (if there is a palpable lump, biopsy pathology suggests) interstitial chronic cell infiltration. At the same time, the special staining of immunohistochemistry is negative [anti-acid, mucicarmine, PAS, fungi (FISH), TB (FISH), methenamine silver], and the possibility of infection with fungi, Mycobacterium tuberculosis or other rod bacteria is ruled out via DNA sequencing using fresh tissue taken from IGM lesions; measurable lesions (mainly low echo lesions detectable by breast ultrasound).

[Exclusion Criteria]

1. Related to subjects:

   Pregnant, breast-feeding, or women planning to have children within 3 years; informed consent does not meet the requirements (if not the patient herself, authorization consent form is missing).
2. Relevant to the disease:

   Core-needle biopsied pathology suggests inflammation caused by pathogens such as tuberculosis or other bacteria, or any item tested positive in the above immunohistochemistry; lung (HR) CT suggests that tuberculosis or tumor cannot be ruled out; Misdiagnosis; No testing records available; No revisit records available.
3. Exclusion criteria related to concomitant medication:

Unable to conduct an efficacy evaluation due to the use of other potential therapeutic drugs, such as glucocorticoids or antituberculosis drugs; Confirmed malignant tumors, those under treatment or after treatment; With severe complications such as cardiac or pulmonary insufficiency, severe cerebral infarction, etc., unable to tolerate treatment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Until progression or recurrence, assessed up to approximately 24 months post-intervention
  Objective response rate (ORR) was defined as the sum of complete response rate (CR) and partial response rate (PR). The largest IGM lesion was evaluated using breast ultrasound (BUS) according to RECIST v1.1 in two dimensions: length ("LGH" in cm) and height ("HGT" in cm). CR was defined as the complete resolution of target lesion confirmed by both physical examination (PE) and BUS, complete healing of skin ulcerations and sinuses, and normalization of 12 inflammatory biomarkers. PR required ≥50% reduction in abnormal inflammatory markers accompanied by at least one of the following criteria: (1) clinical improvement in erythema, edema, local hyperthermia, or pain; (2) ≥50% reduction in LGH or HGT measured by BUS; or (3) ≥75% healing of skin ulcerations and sinuses.

SECONDARY OUTCOMES:
12-month recurrence rate | Until progression, assessed up to approximately 24 months post-intervention
  Relapse rate of IGM within 12 months after discontinuation of baricitinib when achiving CR, decreasing of 12 inflammation markers involving IL1β/IL2/IL4/IL6/IL8/IL10/IL17α/IL12P70/IFNα/IFNγ/TNFα.
Toxicity and side effects | Up to follow-up period, approximately 24 months post-intervention
  Occurrence of adverse events (AEs) after baricitinib administered orally according to NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Wei, Doctor, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China